CLINICAL TRIAL: NCT00797563
Title: Clinical Evaluation of the Apollo Blood Glucose Monitoring System With Capillary and Venous Blood [Commercial Name is CONTOUR® USB]
Brief Title: Evaluation of a New Blood Glucose Meter System With Capillary and Venous Blood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-2008-17
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Results first posted 2009-12-22 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects with diabetes (Other): Subjects with diabetes use a new blood glucose monitoring system (BGMS) Apollo Blood Glucose Monitoring System with capillary blood; healthcare professionals use the new BGMS with subject capillary and venous blood.
  Interventions: Device: Apollo Blood Glucose Monitoring System

INTERVENTIONS:
Device: Apollo Blood Glucose Monitoring System — Subjects with diabetes use a new blood glucose monitoring system with capillary blood; healthcare professionals use the new blood glucose monitoring system with subject capillary and venous blood. All results are compared to a laboratory glucose method - Yellow Springs Instrument (YSI).
  Other Names: CONTOUR® USB

SUMMARY:
The purpose of the study was to evaluate the performance of the meter system in the hands of subjects and healthcare professionals (HCPs). It also evaluated the product user guides in the hands of untrained subjects.

DETAILED DESCRIPTION:
The study evaluated the performance of the blood glucose meter system (BGMS) compared to a laboratory glucose method. Subjects and healthcare professionals tested subject capillary blood and healthcare professionals tested subject venous blood. Two meter configurations were evaluated. The study evaluated the acceptability of product labeling in enabling subjects to perform blood glucose testing with the new meter system and for using meter features. Subjects and healthcare professionals provided feedback about the BGMS and its features.

ELIGIBILITY:
Inclusion Criteria:

* Have type 1 or type 2 diabetes
* Be > 18, < 76 year of age at time of consent, with approximately 50% (+10%)being less than 55 years of age
* Be willing to complete all study procedures
* Be routinely testing their blood sugar at home (at least once per day)
* Be able to speak, read, and understand English and understand the Informed Consent document
* Be able to read the labeling instructions

Exclusion Criteria:

* Minors < 18 years of age and adults > 75 years of age
* Pregnancy
* Physical (dexterity), visual, or neurological impairments that would make the person unable to perform testing with the BGMS
* Disorders in the fingertip lancing areas
* Acute or chronic infections, particularly skin infections
* Infection with a blood borne pathogen
* Taking prescription anti-coagulants or having clotting problems that may prolong bleeding. Taking aspirin daily (81 mg or 325 mg) is not reason for exclusion
* Hemophilia or any other bleeding disorder
* Having a condition which, in the opinion of the Principal Investigator or designee, would put the person at risk or seriously compromise the integrity of the study
* Working for a competitive medical device company

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2008-11; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joy Frank, RN, Principal Investigator — Consumer Product Testing Co., Inc.
Locations (1):
- Consumer Product Testing Co., Inc., Fairfield, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With Diabetes: Subjects with diabetes use a new blood glucose monitoring system (BGMS) with capillary blood; healthcare professionals use the new BGMS with subject capillary and venous blood.
Period: Overall Study
Arm/Group | Subjects With Diabetes
Started | 102 (number of subjects)
Completed | 101
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Subjects With Diabetes
Number analyzed (Participants) | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 70
  >=65 years | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 41
Region of Enrollment [Number; unit: participants]
  United States | 102

OUTCOME MEASURES:

1. Primary Outcome: Number of Capillary and Venous Results Within +/- 15mg/dL or +/- 20% of Laboratory Glucose Method
Description: Subjects with diabetes and healthcare professionals (HCPs) used a new blood glucose monitoring system (BGMS) with subject capillary blood. HCPs used the new bgms with subject venous blood. All results were compared to a lab glucose method. The BGMS has programmed algorithms to provide results equivalent to either serum/plasma or whole blood glucose methods. Number of results were obtained by combining results from three lots of Contour Blood Glucose strips.
Time Frame: One hour
Population: One subject had a non-serious, non-device related anticipated adverse event (a low blood glucose concentration). The subject was treated and discontinued the study.
  The tube collected for the capillary lab glucose assay from one subject was lost in processing, so 100 capillary and 101 venous samples were compared with the lab method.
Measure: Number; unit: number of blood glucose (BG) results
Arm/Group | Subjects With Diabetes
Number analyzed (Participants) | 101
number of blood glucose (BG) results
  Subjects: Capillary Plasma (n=300) | 273
  HCPs: Capillary Plasma (n=300) | 274
  Subjects: Capillary Whole Blood (n=300) | 280
  HCPs: Capillary Whole Blood (n=299) | 273
  HCPs: Venous Plasma (n=605) | 597
  HCPs: Venous Whole Blood (n=606) | 603

2. Secondary Outcome: Percentage of Participants Rated as <=3 (Labeling Comprehension)
Description: Study staff rated participants on their success at performing BG testing and Autolog feature after reading product labeling. The rating scale was:
  1. Successful
  2. Successful after being referred to user instructions
  3. Successful with verbal assistance or review of part of user instructions (Similar to review of a specific function during a Customer Service call.)
  4. Unsuccessful (Incorrectly performed part of the testing regimen or required intervention by study staff.)
Time Frame: One hour
Population: per protocol
Measure: Number; unit: percent of participants
Arm/Group | Subjects With Diabetes
Number analyzed (Participants) | 102
percent of participants
  Perform BG measurement (102/102) | 100
  Select Before/After Meal(Autolog feature) (99/102) | 97

3. Secondary Outcome: Number of Partipants Who Gave These Ratings for Overall Testing Experience With This Meter
Description: Subjects completed a questionnaire rating their overall experience with the Apollo Blood Glucose Monitoring System (User feedback on the system). The rating scale was 0 (Unacceptable) to 4 (Excellent).
Time Frame: One hour
Measure: Number; unit: number of participants
Arm/Group | Subjects With Diabetes
Number analyzed (Participants) | 101
number of participants
  4 Excellent | 68
  3 Very Good | 22
  2 Good | 11
  1 Poor | 0
  0 Unacceptable | 0

ADVERSE EVENTS:
Arm/Group | Subjects With Diabetes
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less